CLINICAL TRIAL: NCT00400803
Title: Phase II Study of Biweekly Carboplatin and Gemcitabine With Bevacizumab as 1st Line Treatment in Patients With Advanced, Inoperable Stage IIIb/IV NSCLC
Brief Title: Carboplatin and Gemcitabine With Bevacizumab Every 2 Weeks for Stage IIIb/IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007UC021; HHH2L06 (Other: Hubert H. Humphrey Cancer Center); AVF3982s (Other: Genentech, Inc.); B9E-US-X463 (Other: Eli Lilly)
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Gemcitabine; Carboplatin; Bevacizumab; Biological therapy; Drug therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Stage IIIb/IV Non-Small Cell Lung Cancer (Experimental): Patients treated with Gemcitabine 2000mg/m^2 intravenously (IV) over 30 minutes, followed by Carboplatin AUC= 3 IV over 30 minutes and Bevacizumab 10 mg/kg IV over 90 minutes 1st infusion, 60 minutes 2nd infusion and 30 minutes for the following infusions. Cycles will be repeated every 2 weeks for a maximum of 6 cycles of therapy. Bevacizumab will continue to be given until disease progression.
  Interventions: Drug: Gemcitabine, Carboplatin, Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine, Carboplatin, Bevacizumab — Patients will be treated with Gemcitabine 2000mg/m^2 intravenously (IV) over 30 minutes, followed by Carboplatin AUC= 3 IV over 30 minutes and Bevacizumab 10 mg/kg IV over 90 minutes 1st infusion, 60 minutes 2nd infusion and 30 minutes for the following infusions. Cycles will be repeated every 2 weeks for a maximum of 6 cycles of therapy. Bevacizumab will continue to be given until disease progression.
  Other Names: Gemzar, Carboplatin, Avastin

SUMMARY:
The purpose of this study is to determine whether treatment with carboplatin and gemcitabine combined with bevacizumab every two weeks will provide increased survival.

DETAILED DESCRIPTION:
Treatment with Carboplatin and gemcitabine is one of the most active combination therapies used for first-line therapy of NSCLC. The optimum schedule for administration of carboplatin and gemcitabine is currently unknown.

The addition of bevacizumab to another comparable platinum combination showed an overall survival advantage and a significantly greater response rate and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC) EXCEPT squamous cell carcinoma or predominantly squamous. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present in which case the patient is ineligible. (Sputum cytology alone is not acceptable)
* Must have disease that is not curative by standard methods.
* Prior adjuvant systemic chemotherapy, immunotherapy, or biological therapy is allowed, except for prior use of bevacizumab. If gemcitabine was used, more than six months must have elapsed between completion of adjuvant therapy and disease progression. Patient must be at least 14 days from previous systemic therapy (at least 30 days for investigational agents) and have recovered from the acute toxic effects of the treatment as determined by the treating physician prior to study registration. Prior therapy other than adjuvant therapy is not allowed.
* Prior radiation therapy must be completed at least 14 days of study registration and subjects must fully recover from acute toxicities as determined by the treating physician. Prior radiation to > 25% of bone marrow is not allowed. Prior radiation therapy to the whole pelvis is not allowed.
* Disease status must be measurable or non-measurable as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* ECOG Performance status of 0 or 1
* Age 18 years or greater
* Adequate organ function within 14 days of study registration including the following:

  * Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, hemoglobin ≥ 9 g/dL
  * Hepatic: bilirubin ≤ 1.5 times the upper limit of normal (× ULN), alkaline phosphatase (ALP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 × ULN (ALP, AST, and ALT ≤ 5 × ULN is acceptable if liver has tumor involvement)
  * Renal: Adequate renal function as evidenced by creatinine clearance of > 50ml/min, estimated by the Cockcroft-Gault equation or urine dipstick for proteinuria < 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
  * Coagulation: INR < 1.5, PTT < the upper limits of normal (ULN) unless stable on therapeutic anticoagulation at study entry. The addition of anticoagulants after study start is not allowed.
* Women of childbearing potential and sexually active males are required to use an effective method of contraception (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicidal, condom with spermicidal, or abstinence) during the study and for 3 months after the last dose of study drug.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Intrathoracic lung carcinoma of squamous cell histology. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is acceptable for inclusion. Subjects with extrathoracic-only squamous cell NSCLC are eligible. Subjects with only peripheral lung lesions of any NSCLC histology will also be eligible. A peripheral lesion is defined as a lesion in which the epicenter of the tumor is < 2 cm from the costal or diaphragmatic pleura in a three-dimensional orientation based on each lobe of the lung and is > 2 cm from the trachea, main and lobar bronchi.
* Pregnant (positive pregnancy test within 14 days of study enrollment) or breast-feeding. Gemcitabine and carboplatin are pregnancy category D - clear evidence of risk in pregnancy; bevacizumab is pregnancy category C - risk in pregnancy cannot be ruled out. Pregnancy testing is not required for post-menopausal (defined as absence of menses for the preceding 24 consecutive months) or surgically sterilized women.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Clinically significant peripheral vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy in the absence of therapeutic anticoagulation
* Current or recent (within 10 days of enrollment) use of aspirin (>325 mg/day) or chronic use of other NSAIDs known to inhibit platelet function Treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal)
* Requiring therapeutic anticoagulation
* Current, ongoing treatment with full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin)
* History of thrombotic or hemorrhagic disorders
* T4 tumors with invasion of the heart or great vessels
* Presence or history of central nervous system or brain metastases, except for treated brain metastases. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI/CT) during the screening period. Anticonvulsants are allowed, providing the subject is on a stable dose. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Subjects with CNS metastases treated by radiotherapy within 28 days of Day 1 will be excluded. Subjects treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* History of another malignancy other than NSCLC except in situ carcinoma of the cervix; adequately treated nonmelanomatous carcinoma of the skin; low grade (Gleason score ≤ 6) localized prostate cancer or other prior malignancy treated at least 2 years previously with no evidence of recurrence
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to treatment start, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to treatment start
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to treatment start
* Serious, non-healing wound, ulcer, or bone fracture, or the presence of a serious active infection
* History of hemoptysis defined as bright red blood of 1/2 teaspoon or more in the previous 1 month before enrollment
* Patients with known hypersensitivity to any of the components of carboplatin, gemcitabine or bevacizumab.
* Known HIV or Hepatitis B or C (active, previously treated or both)
* Inability to comply with study and/or follow-up procedures
* Life expectancy < 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kumar, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Hubert H. Humphrey Cancer Center, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota

REFERENCES:
- [Derived] Dudek AZ, Kumar P, H Thaw SS, Cao Q, Pawloski P, Larson T. Phase II study of biweekly carboplatin, gemcitabine, and bevacizumab as first-line treatment in patients with stage IIIB/IV NSCLC. Am J Clin Oncol. 2014 Apr;37(2):140-3. doi: 10.1097/COC.0b013e31826b9e12. PMID 23111363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 Patients with stage IIIb/IV non-small cell lung cancer were recruited at two institutions in Minnesota: Masonic Cancer Center at University of Minnesota and North Memorial Research Center (Hubert H. Humphrey Cancer Center).
Pre-assignment Details: Outcome data analysis is only available for 35 of 38 patients in database. Three patients are excluded: 1 never enrolled, 1 has no record of treatment and fup, 1 has no treatment fup.
Groups:
- Intent To Treat - Lung Cancer Patients: Patients with Stage III-IV non-small cell lung cancer treated with Gemcitabine 2000mg/m^2 intravenously (IV) over 30 minutes, followed by Carboplatin AUC= 3 IV over 30 minutes and Bevacizumab 10 mg/kg IV over 90 minutes 1st infusion, 60 minutes 2nd infusion and 30 minutes for the following infusions. Cycles will be repeated every 2 weeks for a maximum of 6 cycles of therapy. Bevacizumab will continue to be given until disease progression.
Period: Overall Study
Arm/Group | Intent To Treat - Lung Cancer Patients
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent To Treat - Lung Cancer Patients
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 65 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression (progression free survival)is defined as the time from the start of treatment until first documented sign of disease progression or death due to any cause. For subjects who do not progress, time to progression will be censored at the time of last tumor assessment.
Time Frame: From Enrollment Through 2 Years
Measure: Mean (Standard Error); unit: Months
Arm/Group | Intent To Treat - Lung Cancer Patients
Number analyzed (Participants) | 35
Months | 3.1 (0.4) [79 to 100]

2. Secondary Outcome: Best Overall Response by Cycle
Description: Number of patients and their best response recorded from the state of treatment until disease progression. Response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST): Complete Response-disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that did not meet above criteria.
Time Frame: After Cycle 4, Cycle 6 and Cycle 7 of Therapy
Population: For subjects who show a response, duration of response is defined to be the time from first documented evidence of response until the first documented sign of disease progression or death due to any cause. For subjects who do not progress or die, duration of response will be censored at the time of last tumor assessment. 5 patients = missing data.
Measure: Number; unit: Participants
Groups:
- Intent To Treat - Lung Cancer Patients: Patients with Stage III-IV non-small cell lung cancer treated with Gemcitabine, Carboplatin and Avastin IV every 14 days.
- Partial Response: At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter. To be assigned a status of partial response, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met.
- Stable Disease: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease. To be assigned a status of stable disease, measurements must have met the stable disease criteria at least once after study entry at a minimum interval.
- Progressive Disease: At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Arm/Group | Intent To Treat - Lung Cancer Patients | Partial Response | Stable Disease | Progressive Disease
Number analyzed (Participants) | 35 | 19 | 10 | 6
Participants
  Cycle 1 | 1 | 0 | 0 | 1
  Cycle 2 | 1 | 0 | 0 | 1
  Cycle 3 | 3 | 0 | 2 | 1
  Cycle 4 | 24 | 15 | 6 | 3
  Cycle 5 | 0 | 0 | 0 | 0
  Cycle 6 | 2 | 2 | 0 | 0
  Cycle 7 | 4 | 2 | 2 | 0

3. Secondary Outcome: Duration of Response
Description: For subjects who show a response, duration of response is defined to be the time from first documented evidence of response(30% decrease or complete disappearance of tumor) until the first documented sign of disease progression or death due to any cause. For subjects who do not progress or die, duration of response will be censored at the time of last tumor assessment.
Time Frame: From Enrollment through Date of First Documented Disease Progression or Date of Death From Any Cause, Whichever Came First, Up to 100 Months
Measure: Median (Full Range); unit: Days
Arm/Group | Intent To Treat - Lung Cancer Patients
Number analyzed (Participants) | 35
Days | 105 [4 to 451]

4. Secondary Outcome: Overall Survival Time
Description: Overall survival is defined as the time from the start of treatment until death due to whatever cause. For subjects alive at study completion, time to death will be censored at the time of last contact.
Time Frame: Baseline to Death
Measure: Mean (Standard Error); unit: Months
Arm/Group | Intent To Treat - Lung Cancer Patients
Number analyzed (Participants) | 35
Months | 14.3 (1.3)

5. Secondary Outcome: Time to Best Response
Description: Time to best response is defined as the time from the start of treatment until first documented evidence of tumor response (30% decrease or complete disappearance of tumor). For subjects who do not show a tumor response, the time will be censored at the time of last contact.
Time Frame: From Enrollment to First Tumor Response
Measure: Median (Full Range); unit: Days
Arm/Group | Intent To Treat - Lung Cancer Patients
Number analyzed (Participants) | 35
Days | 72 [42 to 748]

ADVERSE EVENTS:
Arm/Group | Intent To Treat - Lung Cancer Patients
Serious Adverse Events (participants affected / at risk) | 17/38
Other Adverse Events (participants affected / at risk) | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent To Treat - Lung Cancer Patients (N=38)
Ataxia (Nervous system disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Bilateral hearing loss (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Headache (General disorders) | 2 (2)
Hemorrhage, pulmonary (Reproductive system and breast disorders) | 1 (2)
Hypertension (Cardiac disorders) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (General disorders) | 1 (1)
Neutropenia (Infections and infestations) | 1 (1)
Pain, musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 4 (4)
Sensory neuropathy (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (2)
Thrombocytopenia (bruising) (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent To Treat - Lung Cancer Patients (N=38)
Allergy/immunology (Immune system disorders) | 3 (3)
Auditory/Ear (Ear and labyrinth disorders) | 3 (3)
Blood/bone marrow (Blood and lymphatic system disorders) | 6 (12)
Cardiac general (Cardiac disorders) | 12 (13)
Constitutional symptoms (General disorders) | 24 (48)
Dermatology/skin (Skin and subcutaneous tissue disorders) | 8 (18)
Endocrine (Endocrine disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 27 (105)
Hemorrhage/bleeding (Blood and lymphatic system disorders) | 2 (3)
Infection (Infections and infestations) | 8 (10)
Lymphatics (Immune system disorders) | 6 (9)
Metabolic/laboratory (Metabolism and nutrition disorders) | 7 (13)
Musculoskeletal/soft tissue (Musculoskeletal and connective tissue disorders) | 5 (7)
Neurology (Nervous system disorders) | 12 (20)
Ocular/visual (Eye disorders) | 8 (9)
Pain (General disorders) | 23 (68)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 22 (43)
Renal/genitourinary (Renal and urinary disorders) | 4 (4)
Syndromes (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Outcome data is available for 35 (of 38) patients only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes